CLINICAL TRIAL: NCT02859246
Title: Mucinex® for Treatment of Filamentary Keratitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Reza Dana, MD, Reza Dana, MD, MPH, MSc, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-044H
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Filamentary Keratitis
MeSH Terms: interventions — Acetylcysteine; Guaifenesin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mucinex (Other): 600 mg of Mucinex 2 times a day.
  Interventions: Drug: Mucinex®

INTERVENTIONS:
Drug: Mucinex® — Mucinex®
  Other Names: Guaifenesin

SUMMARY:
It is a pilot study aimed to determine if oral Mucinex® is effective in reducing the amount of corneal filaments and improving symptomology in subjects with filamentary keratitis.

DETAILED DESCRIPTION:
The study is aimed to determine if oral administration of Mucinex® is effective in reducing the amount of corneal filaments and improving symptomology in subjects with filamentary keratitis. Subjects will be instructed to take 600 mg tablets of extended release Mucinex® twice a day (total dose is 1.2 g/day) for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with filamentary keratitis
* 18 years and older

Exclusion Criteria:

* Active ocular surface infection of any type
* Recent ocular surgery (<30 days) history of nephrolithiasis as Mucinex® has been associated in rare cases of development of kidney stones
* Schirmer's test<3mm
* History of hypersensitivity to Mucinex®
* Concurrent eye disease requiring immediate initiation of a new treatment (e.g. topical steroids) restriction for water intake can exacerbate the risk of nephrolithiasis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Dana, M.D,MPH,M.Sc, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://doi.org/10.1016/j.jtos.2019.03.008

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mucinex
Started | 15 (15 subjects were enrolled into study)
Completed | 10 (10 subjects completed the study)
Not Completed | 5
Not completed — Screen fails | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All the subjects received Mucinex
Arm/Group | Mucinex
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 63.7 [46 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Number of Corneal Filaments in both eyes [Mean (Standard Deviation); unit: number of corneal filaments] | 2.1 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Corneal Filaments
Description: Change was calculated as the value after receiving treatment with guaifenesin for 4 weeks minus the value at baseline.
Time Frame: baseline (day 1) and week 4
Measure: Mean (Standard Deviation); unit: corneal filaments
Arm/Group | Mucinex
Number analyzed (Participants) | 10
corneal filaments
  number of Corneal filaments at baseline | 5.8 (2.9)
  number of Corneal filaments at week 4 | 2.1 (2.2)
Statistical Analysis 1: Comparison: Mucinex; Test type: Superiority; p < 0.04, Wilcoxon (Mann-Whitney) — A two tail P value of less than 0.05 was considered statistically significant

2. Secondary Outcome: Change in OSDI Score
Description: Change was calculated as the value after receiving treatment with guaifenesin for 4 weeks minus the value at baseline.
  Total score ranges from 0-100. Lower OSDI scores means subjects are experiencing low ocular discomfort. High OSDI scores means subjects are experiencing high ocular discomfort.
Time Frame: baseline (day 1) and week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mucinex
Number analyzed (Participants) | 10
score on a scale
  OSDI score at baseline | 55.6 (25.0)
  OSDI score at week 4 | 46.1 (30.9)
Statistical Analysis 1: Comparison: Mucinex; Test type: Superiority; p < 0.2, Wilcoxon (Mann-Whitney) — A two tail P value of less than 0.05 was considered statistically significant

ADVERSE EVENTS:
Time Frame: From study start following enrollment to study completion (4 weeks).
Description: All the subjects once enrolled into study were followed till they completed their week 4 follow-up visit and were asked about any AE. The PI's contact information was listed on ICF for the subjects to call in course of any AE.
Groups:
- Mucinex (Intervetiion): 600 mg of Mucinex, 2 times a day, for 4 weeks.
Arm/Group | Mucinex (Intervetiion)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT02859246/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT02859246/SAP_001.pdf